CLINICAL TRIAL: NCT04836169
Title: Phase 1: Randomized Evaluation of a System to Deliver Mobile Cognitive Behavioral Therapy to Lower Pain Catastrophizing Scores
Brief Title: Phase 1: Randomized Evaluation of a System to Deliver Mobile Cognitive Behavioral Therapy
Acronym: P1RESPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: InCaveo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InCaveoDanielandDaniel2021
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative; Analgesics, Opioid
Keywords: pain
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- InCaveo EOA System (Experimental): InCaveo EOA System (including integrated CBT but without tapering) group
  Interventions: Device: InCaveo's EOA system with integrated mobile CBT
- Control Group-usual care with pill bottles (No Intervention): UCPB group-usual care with pill bottles

INTERVENTIONS:
Device: InCaveo's EOA system with integrated mobile CBT — integrated pain management therapeutic and tapering system including a software apt that manages and tracks patient-reported outcomes, including pain levels, medication use, quality of life
  Arms: InCaveo EOA System

SUMMARY:
The clinical study described in this Clinical Investigation Plan (CIP) will be completed in two stages, Phase I and Phase II. The results of Phase I will confirm patient use of InCaveo's EOA system with integrated mobile CBT but without tapering to improve The Pain Catastrophizing Scale (PCS) scores, and secondarily scores on the VNS pain scale, the Tampa Scale of Kinesiophobia (TSK), and patient satisfaction scores in the subacute period (defined as 2 weeks to 3 months post TKR). Statistically significant positive results on the Pain Catastrophizing Scale (PCS) will trigger phase 2. Phase 1 will also inform the detailed conditions and patient management algorithms for Phase II.

DETAILED DESCRIPTION:
The InCaveo End Opioid Addiction (EOA) System is an integrated pain management therapeutic and opioid tapering system providing alternate treatment options via self-service Cognitive Behavior Therapy (CBT) built into a mobile software app, patient medication usage, and tracking of patient PROs. It is designed to be used alongside Usual Standard of Care using Pill Bottles or to simplify, Usual Care with Pill Bottles (UCPB) treatment practices. The InCaveo EOA System is designed to improve a set of patient outcome measures, primarily Pain Catastrophizing Scale (PCS) and secondarily the Visual Numeric Pain (VNS), Kinesiophobia (TSK) and satisfaction scores while facilitating the ability of patients to taper off their pain medication faster than through the use of USPB in the management of post-operative pain. In order to reduce confounding variables, the study will focus on pain management following a single surgical procedure: Total Knee Replacement (TKR) surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a Pain Catastrophizing Score >16
2. 55 years of age and older.
3. English speaking.
4. Has a smartphone (iPhone).
5. Able to swallow oral medications.
6. No continuous daily opioid as defined as more than 15 days in the 30 days before surgery.
7. Undergoing TKR surgery.
8. Patients who are willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Diagnosed with Opioid Use Disorder (OUD).
2. Actively using illicit drugs.
3. Allergy to opioids
4. Older than 85 years

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale (PCS) | 60 days
  A measure of the extent of catastrophizing

CONTACTS AND LOCATIONS:
Overall Officials: Hoyman Hong, MD, Principal Investigator — InCaveo

IPD SHARING:
Plan to Share IPD: No